CLINICAL TRIAL: NCT06057623
Title: Type 2 Diabetes Mellitus Influence on Patients With Heart Failure With Preserved Ejection Fraction in Neuromuscular Fatigue and Exercise Capacity
Brief Title: Neuromuscular Fatigue and Exercise Capacity in Patients With Type 2 Diabetes Mellitus and HFpEF
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Other Study IDs: Ics Maugeri CE 2756
Record Dates: First submitted 2023-06-21; First posted 2023-09-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus, Type 2; Heart Failure Preserved Ejection Fraction
Keywords: Heart failure preserved ejection fraction; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Heart Failure, Diastolic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: - Group 1: HFpEF patients with diabetes mellitus (HF-T2DM): patients with a diagnosis of diabetes mellitus in optimized drug therapy, documented by values of glycated hemoglobin (HbA1c) between 6% and 9%
  Interventions: Other: Evaluation of central and peripheral neuromuscular fatigue
- Group 2: - Group 2: HFpEF without diabetes mellitus (HF-NotT2DM): patients with HF in absence of diabetes evidenced by values of glycated hemoglobin (HbA1c) < 6.0%
  Interventions: Other: Evaluation of central and peripheral neuromuscular fatigue

INTERVENTIONS:
Other: Evaluation of central and peripheral neuromuscular fatigue — To define peripheral and central component of fatigue, the investigators will test, before, during and after the fatigue task, the force produced during a Maximal Voluntary Contraction (MVC) and the force produced by the electrically evoked Resting Twitch (RT) produced, at rest, 5 seconds after the MVC.

SUMMARY:
An important feature of patients with HFpEF is impaired exercise tolerance, resulting in worsening and reduced quality of life. Studies in the literature on patients with HFpEF suggest that the limited transport of oxygen to the muscles can be one factor leading to the early development of fatigue during physical activity and reduced effort tolerance. A recent study also shows that patients with HFpEF have an increased susceptibility to both central and peripheral fatigue, suggesting that neuromuscular fatigue may be one of the main mechanisms limiting exercise in this population.

Type 2 diabetes mellitus (T2DM), which affects 90-95% of diabetic patients, is a comorbidity of particular interest in heart failure (HF). In T2DM, as in HF, some observed an altered energy metabolism of the muscle and a shift in the type of muscle fibers. Hyperglycemia influences neuromuscular function and appeared to be one of the major causes of oxidative stress by affecting the intrinsic properties of the muscle (mitochondrial activity and function, myofilaments) related to the expression of force. The impact of diabetes on neuromuscular function is also linked to long-term complications such as diabetic peripheral neuropathy involving impairment of motor nerve conduction and vascular complications. This opens up a rather complex picture suggesting that T2DM in patients with HF could contribute to a further decline in muscle strength by further reducing the aerobic capacity of these patients.

It seems, there are currently no studies in the literature evaluating how much the coexistence of T2DM impacts neuromuscular fatigue and strength in patients with HF. Thus, the primary aim of this study will be to evaluate the differences in central and peripheral neuromuscular fatigue - determined by a submaximal exercise protocol with intermittent isometric contractions - in two groups of patients with heart failure with preserved ejection fraction with or without type 2 diabetes mellitus. Secondary outcomes will be related to the investigation of the differences in NO-mediated vascular function induced by a single passive movement of the leg, in the energy cost of walking, and in muscle oxygenation between the two groups.

DETAILED DESCRIPTION:
The progressive aging of the population of industrialized countries is accompanied by a dramatic increase in the prevalence of chronic diseases. Heart Failure (HF) is one of the major public health problems, with a high incidence of health care costs. In the general population, HF has a prevalence of approximately 1-2% of adults and rises to 10% in the population over 70 years of age.

Heart failure is defined as "the inability of the heart to supply blood adequately to meet the needs of the body, or the ability to do so only at the cost of increased ventricular pressures" Heart failure with preserved ejection fraction (HFpEF) is the most common condition in older adults and its prevalence is increasing as the population ages.

An important feature of patients with HFpEF is impaired exercise tolerance, resulting in worsening and reduced quality of life. Although the attention of the researchers has mostly focused on the definition of central pathophysiological and hemodynamic mechanisms, it has been seen how physical training can improve functional capacity through peripheral adaptive mechanisms that have not been yet clarified. Studies in the literature carried out on this type of patient suggest that the limited transport of oxygen to the muscles is one factor that can lead to the early development of fatigue during physical activity and reduced effort tolerance. A recent study also shows that patients with HFpEF have an increased susceptibility to both central and peripheral fatigue, suggesting that neuromuscular fatigue may be one of the main mechanisms limiting exercise in this population.

Type 2 diabetes mellitus (T2DM), which affects 90-95% of diabetic patients, is a co-condition of particular interest in heart failure, considering the large and ongoing increase in risk associated with heart failure among patients with T2DM. In T2DM, as in HF, it is observed an altered energy metabolism of the muscle and a shift in the type of muscle fibers. Furthermore, hyperglycemia influences neuromuscular function and appears to be one of the major causes of oxidative stress by affecting the intrinsic properties of the muscle (mitochondrial activity and function, myofilaments) related to the expression of force. The impact of diabetes on neuromuscular function is also linked to long-term complications such as diabetic peripheral neuropathy involving impairment of motor nerve conduction and vascular complications. This opens up a rather complex picture that suggests that T2DM in patients with HF could contribute to a further decline in muscle strength by further reducing the aerobic capacity of these patients.

Objective of the study

The primary aim of this study will be to evaluate the differences in central and peripheral neuromuscular fatigue - determined by a submaximal exercise protocol with intermittent isometric contractions - in two groups of patients with heart failure with preserved ejection fraction with or without type 2 diabetes mellitus.

Secondary outcomes: to investigate the differences in NO-mediated vascular function induced by a single passive movement of the leg, in the energy cost of walking, and in muscle oxygenation. These assessments will have the purpose of integrating the assessment of fatigue, to identify the underlying causes.

Measures

The cardiologist will evaluate eligibility to the inclusion/exclusion criteria of patients attending the divisional cardiological visit at Istituti Clinici Scientifici Maugeri (Institute of Lumezzane, Italy) and will request the patient the possibility to join the study, proceeding to collect the informed consent and the following clinical and functional measures present in the patient's clinical documentation: circumferences, weight, height, blood tests, 6-minute walking test, echocardiography. These tests are usually in the patient's possession (preparatory to the cardiological check-up). In the absence of blood exams, tests will be prescribed and scheduled before the start of the study protocol. In any case, glycated hemoglobin will be prescribed for non-diabetic patients.

Regarding therapy and in particular, the drug dapagliflozin, which has recently been introduced into the clinical practice of patients with HFrEF with effects on the reduction of cardiovascular events, there are currently no indications for its use in HFpEF.

Enrolled patients will also be provided with a portable metabolimeter (Dynaport MM, McRoberts), which they will be asked to wear for at least 4 consecutive days before entering the laboratory for testing, in order to monitor their home physical activity profile (main outcome measure: daily steps).

Within one month after the visit, the patient will be invited by a dedicated researcher to go to the gym for the study protocol at the Institute of Lumezzane (BS). There, the patient will perform a series of tests.

Sample size

The sample size was calculated using neuromuscular fatigue as the primary outcome by considering the percentage of change in quadriceps MVC after the fatigue task (percentage of change in maximal isometric force expressed in Newtons). Using data from Weavil et al. (2021) who found a pre-post fatigue MVC reduction of 29 ± 12% in the HFpEF (reference group) and in agreement with Senefeld et al. (2020) who evaluated a reduction in MVC in T2DM of 46.1 ± 11.3%. Assuming an alpha significance level of 0.05 (2-sides), a beta error of 80%, and a 1:1 study-to-control ratio, a minimum total sample size of 20 participants (10 per group) is sufficient to detect significant differences.

Statistical analysis

Data will be analyzed using STATA.12 software. The normality of the distribution for continuous physiological variables will be evaluated with the Shapiro-Wilk test. Data will be expressed as mean ± standard deviation for normally distributed measures or as median (interquartile range) for non-normally distributed measures. For normally distributed data, it will be applied the unpaired or paired t-test for between-group and within-group comparisons, respectively. For data that will not follow a normal distribution, and it will be used the Mann-Whitney U test or Wilcoxon signed-rank test for between-group and within-group comparisons, respectively. The χ2 test will be also applied to compare between-group differences in categorical and binary variables. A P-value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Have a diagnosis of heart failure with preserved ejection fraction (>50%, NYHA class II - III)
2. Have an age between 65 and 80 years
3. Be males
4. Have at least one hospitalization for heart failure during the previous 10 years
5. Have a diagnosis of diabetes for no more than 10 years at the time of cardiology examination

Exclusion Criteria:

* 1. Unstable diabetes documented by HbA1c ≥ 9%
* 2. Significant additional valvular heart diseases
* 3. Unstable heart failure
* 4. Presence of a pacemaker or implanted defibrillator (AICD)
* 5. Changes in drug therapy in the previous three months because of clinical instability
* 6. Body mass index (BMI) > 35 and < 20 kg/m2
* 7. Orthopedic limitations that prevent the exercise
* 8. Presence of diagnosis and signs and symptoms of diabetic neuropathy (intensified perception of pain, burning or cold sensation, tingling, pins, and needles, hypo-hypersensitivity to touch)
* 9. Severe deconditioning (patient is confined to home) or vigorous physical activity (sports or similar activity, estimated as more than two hours/day of vigorous exercise)

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — Because of the limited number of HFpEF females attending our Institute, we restricted the study to the male gender only.
Study Population: Old men, with diagnosis of HFpEF and in additional some of them with Diabetes Mellitus Type II
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change of the isometric force | baseline and up to 1400 secs
  The change in maximal isometric force is a measure to estimate the central and peripheral fatigue.
  Assessment maximal isometric contractions (MVC) pre, at midway through the fatigue protocol, 10' post fatigue protocol and 30' after the fatigue protocol. Maximum force reduction expressed in Newtons will be analyzed. Subjects will be seated upright with back support. The hip and knee will be flexed to 90° and the force will be measured by a force transducer. Change in MCV will be calculated as the difference in percentage between the post-pre fatigue task, as follows: (MVCpost - MVCpre) / MVCpre *100, and expressed as percentage.

SECONDARY OUTCOMES:
Nitric oxide-mediated vasodilation | Baseline
  The evaluation of the vascular function will be performed with a Doppler ultrasound at the level of the common femoral artery, in basal conditions and during the application of the Single Passive Leg Movement (sPLM) technique. The sPLM test will be performed on the right common femoral artery, and measurements will be made using a Doppler ultrasound system (Logiq V4-GE, Milwaukee, WI, USA). The sPLM protocol will consist of 60 seconds of baseline data collection at rest, followed by a 1-second passive flexion-extension of the leg. The leg will then be kept fully extended for the remaining 60 seconds after the movement. For each subject the arterial diameter at rest, the blood flow at rest(LBF), the relative changes will be determined (Dpeak). The peak blood flow values, relative changes from rest after leg movement will be calculated second by second. Leg blood flow will be calculated as LBF = Vmeanπ(D/2)^2 x 60.
Change in muscle oxygenation | Up to 12 seconds
  Monitoring of muscle oxygenation will be performed in vivo in terms of mitochondrial function by the Near InfraRed Spectroscopy (NIRS) method, applying a noninvasive probe on the Vastus Lateralis (VL). We will analyze the relative concentration of deoxyhemoglobin (HHb) and oxyhemoglobin (HbO2) in tissues during the fatigue protocol. Total hemoglobin (THb = HHb + HbO2) and Hb difference (Hbdiff = HbO2 - HHb) will be obtained as derived measurements.
Evaluation of the energy cost of walking | Baseline
  The energy cost of walking is a measure that reflects, through the measurement of oxygen consumption, the energy used for all bodily actions during walking. The test to determine the energy cost of walking (CE) will be performed on a treadmill at an auto-selected speed, wearing the COSMED K5 system (COSMED, Italy)). Subjects will perform a stabilization phase in a sitting position for 5 minutes and then stand on a treadmill for 3 minutes. The duration of the test will be approximately 6 minutes or in any case the time necessary to reach and maintain a 1-minute plateau.
  The energy cost of walking (mL/kg*m) will be calculated according to the formula:
  O2cost = [VO2/kg walking - VO2/kg resting]/speed
Evaluation of Angle of the pennation of Vastus Lateralis | Baseline
  We will use ultrasound scanning for the evaluation of the pennation angle (°) of the Vastus lateralis (VL) muscle in order to investigate differences in muscle architecture. We will take images of the VL at 50% of the thigh length, from the greater trochanter to the superior border of the patella. We will acquire images with an ultrasound device equipped with a linear 8-12 MHz transducer. The pennation angle of the LV bundles will be measured as the angle between the muscle bundles of the LV and the deep insertion aponeurosis.
Evaluation of the Volume of Quadriceps | Baseline
  We will calculate thigh and leg volume (cm3) based on leg circumferences (cm) (at three sites: distal, mid, and proximal), thigh and leg length, and skinfold measurements (cm), using the following formula:
  V= (L ⁄ 12 π) (C12 C22 C32) - [ (S - 0,4 ⁄ 2] L [(C1 C2 C3 )⁄ 3]
  where L=length; C1, C2 and C3 are the proximal, middle and distal circumferences, respectively; and S=skin fold thickness of the thigh or lower leg.
  We will measure leg length in cm; and volume in cm3.
Time to Failure (t-lim) | Up to 1400 secs
  We will collect the time, in seconds, at which we will stop the patient during the fatigue task.
  This value will be used for determining the patient's level of fatigue.
Change of maximal Voluntary Activation (VA) | baseline and up to 1400 secs
  Evaluation of the electrically stimulated resting force (Qtpot) and of the maximum voluntary activation (MVA). The electrical stimulation used will consist of single square wave pulses of 0.1 ms duration, delivered by a constant current stimulator (DS7AH, Digitimer). The intensity of the stimulus used will be defined as follows: the current will be progressively increased from 0 mA to the value beyond which there will be no further increase in force and the amplitude of the M wave. The stimulus used for the study will be set at 125% of the intensity required to produce a maximum M wave response. Voluntary activation (VA) was then assessed using the interpolated twitch technique by comparing the force produced during a superimposed twitch on the MVC with the potentiated single twitch delivered 2-s afterwards.
  %VA = (1 - superimposed twitch force / Qtw,pot) · 100
Muscle electromyography | baseline and up to 1400 secs
  We will collect the M wave from the vastus lateralis after supramaximal electrical stimulation. The intensity of the stimulus used will be defined as follows: we will increase the current progressively from 0 mA to the value beyond which there will be no further increase in the amplitude of the M wave. The stimulus used for the study will be set at 125% of the intensity required to produce a maximum M wave response.
Change of Rate of Perceived Exertion | baseline and up to 1400 secs
  Rate of Perceived Exertion (RPE) assesses subjective perception of muscle exertion (peripheral fatigue). It will be evaluated on a scale score from 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Paneroni, PhD, Study Director — Istituti Clinici Scientifici Maugeri
Locations (1):
- Istituti Clinici Scientifici Maugeri IRCCS, Lumezzane, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Senefeld JW, Keenan KG, Ryan KS, D'Astice SE, Negro F, Hunter SK. Greater fatigability and motor unit discharge variability in human type 2 diabetes. Physiol Rep. 2020 Jul;8(13):e14503. doi: 10.14814/phy2.14503. PMID 32633071
- [Background] Weavil JC, Thurston TS, Hureau TJ, Gifford JR, Kithas PA, Broxterman RM, Bledsoe AD, Nativi JN, Richardson RS, Amann M. Heart failure with preserved ejection fraction diminishes peripheral hemodynamics and accelerates exercise-induced neuromuscular fatigue. Am J Physiol Heart Circ Physiol. 2021 Jan 1;320(1):H338-H351. doi: 10.1152/ajpheart.00266.2020. Epub 2020 Nov 8. PMID 33164549